CLINICAL TRIAL: NCT04862871
Title: Enhancing Analgesia in Chronic Pain Through Exercise: Responsivity of Sensory-Motor Networks and Factors That Moderate the Analgesic Response
Brief Title: Enhancing Analgesia in Chronic Pain Through Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Scott Holmes, Research Associate, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-P00034939
Record Dates: First submitted 2021-04-16; First posted 2021-04-28 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Pain; Chronic Widespread Pain; Fibromyalgia
MeSH Terms: conditions — Pain; Chronic Pain; Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Participants will be evaluated in three independent groups (healthy controls, participants who have completed an exercise program, participants who are waiting to complete an exercise program).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Controls (No Intervention): A cohort (n=10) of participants will be recruited who do not have any neurological conditions and are age and sex-matched to participants in Arms 2 and 3.
- Chronic Widespread Pain (No Intervention): A cohort (n=10) of participants who have not yet begun the exercise program and are currently on the waitlist for the exercise program at the PPRC
- Chronic Widespread Pain - Exercise (Active Comparator): A cohort (n=10) of participants who have completed the exercise program at the PPRC. These individuals will be evaluated the day of their last treatment visit
  Interventions: Behavioral: Physical Activity - Pediatric Pain Rehabilitation Center

INTERVENTIONS:
Behavioral: Physical Activity - Pediatric Pain Rehabilitation Center — While admitted to the Pediatric Pain Rehabilitation Center program, patients receive 1-3 hours of individual and group physical therapy 5 times per week and completed a 30-60 minute home exercise program 9 times per week. The median length of stay for the program is 5 weeks. The amount of aerobic exercise prescribed is individualized to each patient and ranged from 10-20 minutes per session. The duration of aerobic exercise prescribed progressed by 5-10 min weekly until the child reached 20-30 minutes. Patients are instructed to reach a moderate to vigorous intensity of exercise (defined at 5-7/10 rate of perceived exertion). The mode of exercise varied dependent on patient ability and interest. Typical modes of exercise included: walking, running, stationary biking, swimming, sports (i.e., soccer, dance), and online aerobic workouts. Patients were prescribed an individualized 30-60 minute discharge home program using the same structure upon completing the program.
  Arms: Chronic Widespread Pain - Exercise

SUMMARY:
Background: Current pain management strategies for pediatric patients are not integrating the analgesic potential of movement-based therapies. To date, experiencing a painful stimulus has been known to disrupt motor activity in an attempt to minimize injury. However, physical activity, even when it increases ongoing pain initially, has been shown to significantly reduce pain symptoms eventually through neuromodulation. In both acute and chronic pain cohorts, exercise protocols and neuromodulation paradigms have produced exercise-related analgesia. Problem: It is not currently understood which brain regions are implicated in exercise-based analgesia and what brain regions moderate this response.

Approach: The investigators intend to provide a physical activity intervention designed to promote exercise-induced analgesia. This intervention will be performed in a group of pediatric subjects with Chronic Widespread Pain Disorder. An exercise (n=10), no exercise (n=10) and healthy control (n=10) group will be recruited. Aims: This study has three aims: (1) To understand how thermal pain sensitivity, pain symptoms and motor performance are impacted in patients with chronic pain after an exercise-based intervention. (2) To evaluate the brain regions involved in a simple motor task as well as how motor activity influences activity in pain regions of the brain. (3) To evaluate the network structure of the brain, with special emphasis on motor and pain regions, in youth with a pain disorder who have undergone an exercise-based intervention. Exercise-based therapy in pediatric subjects with a chronic pain condition is predicted to reduce pain symptom reporting through biasing activity in pain regions during motor performance. Significance: Findings from this investigation will address the clinical side of pain management strategies and provide potential therapeutic targets and feasibility data. The investigators anticipate that findings will show how pain and motor regions of the brain interact at the network level and if this interaction can be modulated through exercise. Findings will also evaluate the brain regions that mediate the analgesic properties of an exercise-based pain therapy and provide future therapeutic targets.

DETAILED DESCRIPTION:
This investigation is aimed at understanding how an exercise program currently performed at the Pediatric Pain Rehabilitation Center (PPRC) at Boston Children's Hospital, designed for individuals with chronic widespread pain is associated with pain relief and how this pain relief relates to changes in the brain. The specific aims/objectives are to explore the following:

Aim 1 - Pain and sensorimotor behavior: To understand how thermal pain sensitivity, pain symptoms and motor performance are impacted in children with chronic pain after an exercise-based intervention. Sensory testing (for Hot & Cold) will be collected using Quantitative Sensory Testing (QST) to establish pain thresholds. To address motor performance, we will perform the Bruininks-Oseretsky Test (BOT) 1 of motor proficiency (examining muscle power, strength, endurance). Pain symptom levels will be evaluated using self-report questionnaires that address fear of pain, pain catastrophizing, and pain symptom load.

Aim 2 - Defining hierarchies during motor performance: To evaluate the brain regions involved in a simple motor task as well as how motor activity influences activity in pain regions. Participants will perform a tapping task within the MRI scanner to evaluate the brain regions that are active during motor control. 2 Functional magnetic resonance images will be processed using dynamic causal modeling (DCM) to evaluate effective connectivity (Figure 2) during task performance. Brain regions evaluated in DCM will be defined by the healthy control cohort.

Aim 3 - Network structure: To evaluate the network structure of the brain, with emphasis on motor and pain regions, in persons with a pain disorder who have undergone an exercise intervention. Graph theory analyses implemented using resting-state functional magnetic resonance imaging will be performed to extract metrics reflecting network efficiency, nodal degree, and nodal centrality. Structural metrics (e.g., cortical thickness and white matter connectivity) will be collected as nuisance variables. Correlation analyses will be performed between network metrics and behavior (fear of pain, pain catastrophizing, motor performance) to evaluate their influence over network reorganization observed from the exercise intervention. Brain regions that define canonical pain and motor networks will be indexed from the healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy participants between the ages of 10 and 24
* Actively on the waitlist for, or having completed the exercise program at the PPRC
* Comprehension of instructions
* Parental consent for minors
* Weight less than 250 lbs - limit of MRI table
* Clinical diagnosis of Chronic Widespread Pain

Exclusion Criteria:

* Preventative medications and opioids
* Metallic implants that will pose harm to the subject (e.g., pacemaker) and/or affect the dat (e.g., braces)
* Significant medical disease (systemic or CNS).
* Active suicidality, psychosis, diagnosed eating disorders, and/or other severe clinically diagnosed neuro-psychiatric conditions
* Pregnant
* Claustrophobia

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in effective connectivity | 8 months
  Difference in effective connectivity between motor and pain regions of the brain between persons who have completed the PPRC intervention and those on the waitlist. Whole-brain effective connectivity will be evaluated and compared between groups that will be age and sex-matched. Effective connectivity will be calculated using dynamic causal modeling and evaluated using a tapping task. Effective connectivity will be calculated from a motor task requiring participants to complete an active (tapping) and rest (no tapping) condition.

SECONDARY OUTCOMES:
Thermal sensitivity | 8 months
  Quantitative sensory testing (QST) will be used to evaluate thermal sensitivity to hot and cold stimulus paradigms. The outcome measure of interest will be participants self-reported pain ratings using a visual analogue scale (VAS) from 0 (minimum - no pain) to 10 (maximum - high pain) at specific levels of thermal sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Holmes, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share individual participant data.